CLINICAL TRIAL: NCT04140318
Title: Efficacy and Safety of Sintilimab and Nab-paclitaxel in Advanced Gastric and Gastro-esophageal Junction Adenocarcinoma Patients With Progression After Fluoropyrimidine or Platinum, a Multi-center, Phase II, Single Arm Trial
Brief Title: Sintilimab and Nab-paclitaxel in Second-line Treatment of Advanced Gastric or Gastro-oesophageal Junction Adenocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Chinese PLA General Hospital (Other); Beijing Friendship Hospital (Other); Beijing Hospital (Other Government)
Responsible Party: Principal Investigator, Aiping Zhou, Prof., Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC2070
Record Dates: First submitted 2019-10-24; First posted 2019-10-25 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Advanced Gastric and Gastro-esophageal Junction Adenocarcinoma
Keywords: second line; PD-1; nab-paclitaxel
MeSH Terms: interventions — sintilimab; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment (Experimental): combination therapy of PD-1 and chemotherapy including: sintilimab 200mg iv, 30-60min, q3w; nab-paclitaxel 125mg/m2, iv, d1,d8, q3w
  Interventions: Drug: sintilimab; Drug: nab-paclitaxel

INTERVENTIONS:
Drug: sintilimab — Sintilimab 200mg, iv, 30-60min, q3w;
Drug: nab-paclitaxel — Nab-paclitaxel: 125 mg/m2 iv d1、d8, q3w

SUMMARY:
To evaluate the efficacy and safety of Sintilimab (PD-1 inhibitor) and nab-paclitaxel in second line treatment of advanced gastric and gastro-esophageal junction adenocarcinoma. This is a prospective, multi-centers, single arm phase II trial with primary objective overall response rate and second objective of safety and other efficacy endpoints.

ELIGIBILITY:
Inclusion Criteria:

* pathological confirmed advanced gastric and gastro-esophageal junction adenocarcinoma;
* progression after first-line treatment of fluoropyrimidine and platinum, allow patients progressed on/within 6 months of neoadjuvant/adjuvant treatment; allow local radiotherapy after 21days later;
* 18-75 years old;
* ECOG: 0 or 1;
* has adequate organ function
* writen ICF;

Exclusion Criteria:

* previous treated with taxanes (including paclitaxel, nab-PTX, lipo-PTX, and docetaxel etc..);
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-CTLA-4 antibody;
* has known active central nervous system metastatases;
* has received a live vaccine within 4 weeks prior to the first dose of study treatment with any acitve autoimmune disease or history of autoimmune disease, including but not limited to the following: hepatititis, pneumonitis, uveitis, colitis (inflammatory bowel disease), hypophysitis, vasculitis, nephritis, hyperthyroidism, and hypothyroidism, except for subjects with vitiligo or resolved childhood asthma/atopy. Asthma that requires intermittent use of bronchodilators or other medical intervention should also be excluded.
* clinically significant cardiovascular and cerebrovascular diseases, including but not limited to severe acute myocardial infarction within 6 months before enrollment, unstable or severe angina, Congestive heart failure (New York heart association (NYHA) class > 2), orventricular arrhythmia which need medical intervention.
* hypertension and unable to be controlled within normal level following treatment of anti-hypertension agents(within 3 months): systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg. coagulation abnormalities (INR > 1.5 or APTT > 1.5×ULN), with bleeding tendency or are receiving thrombolytic or anticoagulant therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-11-15 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
ORR | up to two years

SECONDARY OUTCOMES:
DCR | up to three years
  disease control rate
DOR | up to three years
  duration of response
AE | from first dose to 90days of last dose
  treatment related adverse event
PFS | up to three years
  progression free survival
OS | up to three years
  overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided
The baseline characteristics of patients could be shared to othter researchers per request.